CLINICAL TRIAL: NCT00881777
Title: Radiofrequency Energy Use in Cardiomyopathy and Ventricular Enlargement (RECOVER)
Brief Title: Feasibility Study of Radiofrequency Heating of Cardiac Infarction Scar to Treat Heart Failure
Acronym: RECOVER
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit suitable subjects within a reasonable time period.
Sponsor: CoRepair, Inc. (Industry)
Responsible Party: Andrew J. Ford, Jr. / Director of Clinical Affairs, CoRepair, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-01 Rev. C
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Cardiomyopathy; Ventricular Dysfunction; Heart Disease
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Ventricular Dysfunction; Heart Diseases | interventions — Coronary Artery Bypass; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- RF Heating + CABG (Experimental): Radiofrequency heating of the myocardial infarct scar plus Coronary Artery Bypass Grafting (CABG) surgery
  Interventions: Procedure: Radiofrequency heating of the myocardial infarct scar; Procedure: Coronary Artery Bypass Grafting (CABG) surgery
- CABG Alone (Active Comparator): Coronary Artery Bypass Grafting (CABG) surgery only, without radiofrequency heating of the myocardial infarct scar
  Interventions: Procedure: Coronary Artery Bypass Grafting (CABG) surgery

INTERVENTIONS:
Procedure: Radiofrequency heating of the myocardial infarct scar — Radiofrequency energy is applied to the epicardial surface of the heart using an external generator and a hand-held probe to heat myocardial infarction scar.
  Arms: RF Heating + CABG
Procedure: Coronary Artery Bypass Grafting (CABG) surgery — A standard surgical procedure performed to relieve angina and reduce the risk of death from coronary artery disease. Arteries or veins from elsewhere in the body are grafted to the coronary arteries to bypass atherosclerotic narrowings and improve the blood supply to the coronary circulation supplying the myocardium.

SUMMARY:
The purpose of this study is to examine the safety and potential effectiveness of a new surgical procedure for treating heart failure. The experimental treatment is performed during standard coronary artery bypass graft (CABG) surgery, and applies radiofrequency energy to heat a portion of the damaged heart muscle. The tissue heating reduces the enlarged heart of patients suffering from ischemic heart failure, and may result in the heart pumping blood more efficiently, thereby improving the functional status of the patient.

DETAILED DESCRIPTION:
Heart failure is an important health-care problem, resulting in significant numbers of patients, hospitalizations, and economic costs. The etiology of heart failure is coronary artery disease in approximately two-thirds of cases, and the majority of these patients have experienced prior myocardial infarction. As a consequence of the myocardial infarction, the ventricle undergoes changes in volume and shape, a process referred to as "ventricular remodeling". As the left ventricle enlarges, global systolic function worsens, resulting in heart failure. There are a number of treatment options available to minimize symptoms and somewhat slow disease progression. Unfortunately, even with best conventional drug and device therapies, heart failure patients continue to have high morbidity and mortality rates. The experimental therapy investigated in this study uses a surgical device which employs radiofrequency energy to heat epicardial tissue. The application of heat to a myocardial infarction scar causes it to shrink in size, and correspondingly reduces ventricular volume. The volume reduction may "reverse remodel" the enlarged and dysfunctioning left ventricle to a more normal size and shape. The intent of this clinical study is to evaluate whether radiofrequency heating of the myocardial infarct scar is safe, and determine if the resulting ventricular volume reduction translates into improved clinical and functional outcomes in patients suffering from ischemic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, inclusive
* Symptomatic heart failure (defined as persistent NYHA class II or III during the 3 months prior to enrollment)
* On evidence-based medical therapy for heart failure during the 1 month prior to enrollment
* Referred for elective coronary artery bypass grafting
* Dyskinetic transmural myocardial infarct located in the apical portion of the anterior, lateral, and/or inferior left ventricular wall as determined by transthoracic echocardiography ("transmural" means end-diastolic wall thickness of 4 - 6 mm, inclusive)
* Left ventricular ejection fraction 20 - 45%, inclusive as determined by transthoracic echocardiography
* Left ventricular end-systolic volume index ≥ 60 ml/m2 as determined by transthoracic echocardiography
* 6-minute walk distance over 150 m
* Peak VO2 (ml/kg/min): 10.0 - 20.0 for males and 9.0 - 18.0 for females

Exclusion Criteria:

* Myocardial infarction ≤ 3 months prior to enrollment
* Evidence of calcification within the scar intended to be treated by any imaging modality
* Presence of a coronary stent within the scar intended to be treated
* Evidence of left ventricular thrombus
* Emergent cardiac surgery
* Percutaneous coronary intervention (PCI) ≤ 1 month prior to enrollment or planned following enrollment
* Only for patients undergoing MR (rather than CT) imaging: Contraindications for MRI (current or anticipated during the 6 months following enrollment), such as pacemaker, Automatic Implantable Cardioverter-Defibrillator (AICD), Cardiac Resynchronization Therapy (CRT) device, central nervous system aneurysm clips, Cochlear implant, or metal shrapnel
* Only for patients undergoing MR (rather than CT) imaging: Acute or chronic severe renal insufficiency (i.e. a glomerular filtration rate < 30 ml/min/1.73m2) or acute renal insufficiency of any severity due to hepato-renal syndrome
* Only for patients undergoing MR (rather than CT) imaging: Known allergy or reaction to Gadolinium
* Atrial fibrillation
* Prior cardiac surgery (including coronary artery bypass grafting, valve replacement or repair, aortic root replacement) or anticipated during the 6 months following enrollment
* Major non-cardiac surgery (e.g. knee or hip replacement, laparotomy, carotid endarterectomy, etc.) ≤ 3 months prior to enrollment or planned during the 6 months following enrollment
* Prior heart, kidney, liver, or lung transplantation
* Valvular heart disease requiring replacement or repair (e.g. mitral valve regurgitation ≥ 3+)
* Cardiogenic shock ≤ 72 hours prior to the CABG surgery (defined as need for Intra-Aortic Balloon Pump or requiring intravenous inotropic support)
* Currently needing (or anticipated need for) Left Ventricular Assist Device or other cardiac replacement device
* On active heart transplant list or anticipated need for transplant during the 6 months following enrollment
* Stoke or transient ischemic attack ≤ 3 months prior to enrollment
* Chronic dialysis
* Major infection or sepsis ≤ 72 hours of enrollment (defined as requiring IV antibiotics for > 3 days)
* Endocarditis, myocarditis, or pericarditis
* Co-morbid condition that, in the investigator's opinion, results in the patient's life expectancy being < 180 days
* Evidence of significant blood chemistry abnormalities, including creatinine > 2.5 mg/dl, BUN ≥ 100 mg/dl, liver function tests > 3 times upper limit of normal, Hgb < 10 gm/dl, HCT < 25%, platelet count < 100,000/mm3, or white blood cell count < 3,000/mm3 or > 20,000/mm3
* Females of child-bearing potential without a documented negative pregnancy test within the 14 days prior to enrollment (and prior to the MRI or CT) or who are unwilling to use effective contraception for the duration of this study
* Participation in another investigational device or drug trial
* Unable or unwilling to give Informed Consent
* Unwilling or unlikely to complete the required follow-up
* Any other medical condition that, in the judgment of the investigator, would cause this study to be detrimental to the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular End Diastolic and Systolic Volume Indexes as measured by Cardiac MRI/CT | 6 Months
Occurrence of any of the following: cardiac hemorrhage/rupture, cardiac tamponade, stroke/transient ischemic attack/renal failure, myocardial infarction, sepsis/cardiac-related infection, re-hospitalization for cardiac cause, or all-cause mortality | 6 months

SECONDARY OUTCOMES:
Change in Left Ventricular End Diastolic and Systolic Dimensions, Volumes, and Volume Indexes, and Left Ventricular Ejection Fraction as measured by Cardiac MRI/CT | Peri-operative, 6 and 12 months
Change in New York Heart Association Functional Classification and Canadian Cardiovascular Society Angina Grading Scale | 1, 3, 6, and 12 months
Change in Cardiopulmonary Exercise Stress Test (Peak VO2 and VE/VCO2 slope) | 6 and 12 months
Change in 6-Minute Walk distance | 1, 3, 6, and 12 months
Change in Quality of Life Questionnaire score (Minnesota Living With Heart Failure and EuroQol EQ-5D) | 1, 3, 6, and 12 months
Occurrence of individual primary safety endpoints, heart failure deaths, heart failure hospitalizations, all-cause hospitalizations, days alive out of the hospital, and neurological assessments (NIH Stroke Scale and Mini-Mental Status Exam) | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Sanatorio Italiano, Asunción, Paraguay
- Poland (2):
  - The Cardinal Stefan Wyszynski Institute of Cardiology, Warsaw
  - Silesian Center for Heart Diseases, Zabrze

REFERENCES:
- [Background] Ratcliffe MB, Wallace AW, Teerlink JR, Hong J, Salahieh A, Sung SH, Keung EC, Lee RJ. Radio frequency heating of chronic ovine infarct leads to sustained infarct area and ventricular volume reduction. J Thorac Cardiovasc Surg. 2000 Jun;119(6):1194-204. doi: 10.1067/mtc.2000.105826. PMID 10838539
- [Background] Victal OA, Teerlink JR, Gaxiola E, Wallace AW, Najar S, Camacho DH, Gutierrez A, Herrera G, Zuniga G, Mercado-Rios F, Ratcliffe MB. Left ventricular volume reduction by radiofrequency heating of chronic myocardial infarction in patients with congestive heart failure. Circulation. 2002 Mar 19;105(11):1317-22. doi: 10.1161/hc1102.105566. PMID 11901042